CLINICAL TRIAL: NCT05971537
Title: Clinical Trial on Antibiotic-Lock in Tenckhoff Catheter for Relasping and Repeat Peritonitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alice Ho Miu Ling Nethersole Hospital (Other)
Responsible Party: Principal Investigator, chan ping kwan, Associate Consultant, Department of Medicine, Alice Ho Miu Ling Nethersole Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016.513-T
Record Dates: First submitted 2023-05-23; First posted 2023-08-02 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Peritoneal Dialysis-associated Peritonitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention arm (Active Comparator): in addition to the appropriate IP antibiotics, an antibiotic-lock will be prepared by the same antibiotics. We will follow the suggested data used in hemodialysis catheter for the concentration of different antibiotics to prepare the locking solution The resulting locking solution will be instilled precisely to fill up the Tenckhoff catheter and the transfer set once a day. Prior to that, the existing PD solution is drained out first. As such, a "dry abdomen" is maintained during antibiotic-lock dwelling in the Tenckhoff catheter. This is to ensure the antibiotic-lock solution can be maintained within the catheter lumen for a prolonged period of time After a 6-hour dwell, the antibiotic-lock is drained out and usual PD schedule is resumed. Such a daily application of antibiotic lock shall last until the course of IP antibiotics is completed.
  Interventions: Drug: antibiotic lock
- control arm (Other): In the control arm, appropriate IP antibiotics are to be continued. The dosage and duration of antibiotics will fully follow the recommendation from the latest International Society for Peritoneal Dialysis (ISPD) peritonitis guidelines
  *For the subjects in the control arm who reach the defined primary end-point, they will automatically undergo crossover to the intervention arm to receive standard IP antibiotics together with the intra-catheter antibiotic-lock. They will be followed for another 6 months subsequently.
  Interventions: Drug: conventional IP antibiotics

INTERVENTIONS:
Drug: antibiotic lock — In the intervention arm, in addition to the appropriate IP antibiotics, an antibiotic-lock will be prepared by the same antibiotics. We will follow the suggested data used in hemodialysis catheter for the concentration of different antibiotics to prepare the locking solution . Some commonly used antibiotics for the treatment of PD peritonitis with their suggested concentrations in the antibiotic-lock are quoted as below:
  Cefazolin 10mg/mL Ceftazidime 10mg/mL Vancomycin 10mg/mL Gentamicin 5mg/mL Tienam 50mg/mL
  Arms: intervention arm
Drug: conventional IP antibiotics — In the control arm, appropriate IP antibiotics are to be continued. The dosage and duration of antibiotics will fully follow the recommendation from the latest International Society for Peritoneal Dialysis (ISPD) peritonitis guidelines
  Arms: control arm

SUMMARY:
Biofilm formation is an important cause of catheter-related infection. In hemodialysis, use of an antibiotic-lock has been proven to be effective to manage such a complication with preservation of the central venous catheter. In peritoneal dialysis, while biofilm has been implicated in relapsing and repeat peritonitis, both of which are caused by the identical bacteria as in their preceding peritonitis episode, no adjunctive measure has been proven to be effective to eradicate the biofilm bacteria. As a result, Tenckhoff catheter removal is the only recommended option for the patients suffering from relapsing or repeat peritonitis. In this study, the investigators are going to investigate whether the use of an antibiotic-lock can be useful to eradicate the biofilm in the Tenckhoff catheter to prevent future episodes of peritonitis caused by the same organism.

DETAILED DESCRIPTION:
STUDY OBJECTIVES This study aims to evaluate whether the use of antibiotic-lock in the Tenckhoff catheter can eradicate the biofilm within the catheter lumen, thereby preventing further episodes of relapsing of repeat peritonitis without catheter removal.

METHODS Total 46 patients are to be recruited

When a PD patient, who has an episode of peritonitis treated successfully by IP antibiotics within the preceding 12 weeks, returns to the investigator's unit for peritonitis, the patient will be resumed on the same IP antibiotics treatment as in the last episode, while waiting for the PD effluent culture results. In the investigators' experience, the turnaround time of the microbiology report is usually 3-5 days. During this period, the patient should be closely monitored for the response to the antibiotics. The patient will be eligible for recruitment into this study if the same causative organism is confirmed subsequently. Another scenario is the absence of peritonitis symptoms, including PDE leukocyte count <100/mm3, yet there is a persistent growth of bacteria from the PDE after completion of 2-week antibiotic therapy. These patients are also eligible for study recruitment.

After recruitment, the subject will be randomized into either the intervention arm or the control arm in a 1:1 manner. In the control arm, appropriate IP antibiotics are to be continued. The dosage and duration of antibiotics will fully follow the recommendation from the latest International Society for Peritoneal Dialysis (ISPD) peritonitis guidelines. In the case of persistent bacterial growth from PDE without peritonitis symptoms, IP antibiotics will be extended up to 2 weeks more. In the intervention arm, in addition to the appropriate IP antibiotics, an antibiotic-lock will be prepared by the same antibiotics. The investigators will follow the suggested data used in hemodialysis catheter for the concentration of different antibiotics to prepare the locking solution

All antibiotics are diluted into an appropriate amount of normal saline or water to achieve the desired concentration. The resulting locking solution will be instilled precisely to fill up the Tenckhoff catheter and the transfer set once a day by the renal nurses. Prior to that, the existing PD solution is drained out first. As such, a "dry abdomen" is maintained during antibiotic-lock dwelling in the Tenckhoff catheter. This is to ensure the antibiotic-lock solution can be maintained within the catheter lumen for a prolonged period of time. After a 6-hour dwell, the antibiotic-lock is drained out and usual PD schedule is resumed. Such a daily application of antibiotic lock shall last until the course of IP antibiotics is completed.

RANDOMIZATION Randomization is carried out by drawing a consecutively numbered, sealed, opaque envelope containing a form indicating whether the subject is randomized into the intervention arm or control arm.

STUDY PARAMETERS The patients' demographics, including the age, gender, body mass index, PD vintage, etiology of end-stage renal disease, co-morbidities, together with the previous PD peritonitis history will be retrieved. The causative organisms of the current relapsing or repeat peritonitis are recorded.

After recruitment into the study and the peritonitis episode has been cured successfully, all subjects will be followed for up to 6 months after completion of their IP antibiotics treatment.

TERMINATION OF STUDY The subjects will be out from the trial when they have completed the study, or before the end of the study if their peritonitis is refractory to appropriate IP antibiotics rendering a need of timely Tenckhoff catheter removal, or at anytime the subjects decide to withdraw from the trial.

ELIGIBILITY:
Inclusion Criteria:

* PD patients who suffer from Either relapsing peritonitis (within 4 weeks of completion of antibiotics) or repeat peritonitis (between 4 to 12 weeks of completion of antibiotics), in which the causative organism is confirmed to be identical to the one in the preceding peritonitis episode, or Persistent growth of bacteria from PD effluent (PDE) after completion of standard 2-week antibiotic treatment, despite the resolution of symptoms and PDE leukocyte count <100/mm3
* Age > 18 years old
* informed consent available

Exclusion Criteria:

* Patients who do not respond to the appropriate IP antibiotics, evident by the persistence of peritonitis symptoms in which they should be referred for timely Tenchkoff catheter removal
* Fungal or mycobacterial PD peritonitis
* Co-existing exit site or tunnel tract infection
* The presence of Tenckhoff catheter drainage dysfunction
* <= 3 years old
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
rate of developement of relapsing or repeat peritonitis | 6 month
  Development of relapsing peritonitis (within 4 weeks of completion of antibiotics) or repeat peritonitis (between 4 to 12 weeks of completion of antibiotics) again

SECONDARY OUTCOMES:
rate of development of peritonitis due to same organism, beyond 12 weeks | 6 month
  Development of peritonitis due to the same organism, beyond 12 weeks of completion of antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: ping kwan chan, Principal Investigator — Alice Ho Miu Ling Nethersole Hospital
Locations (1):
- Alice Ho Miu Ling Nethersole Hospital, Tai Po, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li PK, Szeto CC, Piraino B, de Arteaga J, Fan S, Figueiredo AE, Fish DN, Goffin E, Kim YL, Salzer W, Struijk DG, Teitelbaum I, Johnson DW. ISPD Peritonitis Recommendations: 2016 Update on Prevention and Treatment. Perit Dial Int. 2016 Sep 10;36(5):481-508. doi: 10.3747/pdi.2016.00078. Epub 2016 Jun 9. No abstract available. PMID 27282851
- [Background] Justo JA, Bookstaver PB. Antibiotic lock therapy: review of technique and logistical challenges. Infect Drug Resist. 2014 Dec 12;7:343-63. doi: 10.2147/IDR.S51388. eCollection 2014. PMID 25548523
- [Background] Wong SS, Lau WY, Chan PK, Wan CK, Cheng YL. Extended Experience in the Use of Antibiotic Lock for Eradication of Biofilm Bacteria on Tenckhoff Catheter. Perit Dial Int. 2019 Mar-Apr;39(2):187-190. doi: 10.3747/pdi.2018.00098. PMID 30858288